CLINICAL TRIAL: NCT05000268
Title: Examination of The Effects of Telerehabilitation in Painful Healthcare Workers With and Without COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ceyhun Topcuoğlu, Principal Investigator, Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-CT-04
Record Dates: First submitted 2021-08-06; First posted 2021-08-11 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Respiratory Infection
Keywords: COVID-19; telerehabilitation; pain; healthcare workers; progressive myofascial relaxation technique
MeSH Terms: conditions — COVID-19; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups as those with pain after COVID-19 infection and those with pain not related to COVID-19 infection. Both groups will be applied telerehabilitation methods, progressive myofascial relaxation techniques and simple posture correction exercises every other day for 2 weeks. Progressive myofascial relaxation exercises will be asked to do morning and evening while lying in bed. Posture exercises will be required to perform while standing, at least 2 or 3 sets during work.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painful Healthcare Workers with COVID-19 (Active Comparator): Healthcare workers who have had COVID-19 infection in the past and are now in pain without COVID-19 infection
  Interventions: Other: Progressive Myofascial Relaxation Exercise
- Painful Health Care Workers without COVID-19 (Active Comparator): Healthcare workers with past and present pain without COVID-19 infection
  Interventions: Other: Progressive Myofascial Relaxation Exercise

INTERVENTIONS:
Other: Progressive Myofascial Relaxation Exercise — Participants will be given telerehabilitation methods, progressive myofascial relaxation techniques and simple posture correction exercises every other day for 2 weeks. The exercises will be performed as follows:
  * First, focus on creating tension in the body by contracting all your body muscles and feeling the body tension by holding this tight position for 3-5 seconds. Then relax and relax and focus on feeling the relaxed position of the muscles for 10-15 seconds. Then, the same contraction and relaxation movements will be applied in the feet, legs, hips, waist, chest, shoulders, arms and face areas, respectively. They will be asked to do these exercises in the morning and evening while lying in bed.

SUMMARY:
In the literature, there are studies examining the effects of telerehabilitation on individuals who have had COVID-19, but studies examining the effects on healthcare workers who have experienced COVID-19 are insufficient. In this study, which is planned to be done, it is aimed to examine the effects of myofascial relaxation technique on pain and other symptoms through telerehabilitation. The aim of the study is to examine the effects of myofascial relaxation technique applied with the telerehabilitation method on pain level, anxiety, depression, sleep, fatigue and kinesiophobia in healthcare workers with and without COVID-19 infection with pain.

DETAILED DESCRIPTION:
COVID-19 is a disease caused by severe acute coronavirus 2 infection and declared as a pandemic by the World Health Organization on March 11, 2020. In the period from March 11, when the first case was announced in Turkey, to the present day, the total number of cases has exceeded 2.3 million. COVID-19 is mainly transmitted by air droplets, aerosols and direct contact, and asymptomatic carriers are the main reason for rapid spread. While many professional groups are working at home during the pandemic process; the risk of contracting COVID-19 has increased, especially in healthcare workers working in high-risk departments of hospitals where COVID-19 patients are treated.

Along with symptoms such as fever, dry cough and shortness of breath, common musculoskeletal problems such as muscle pain, joint pain and fatigue, anxiety, depression and deterioration in sleep quality have been observed in COVID-19 patients. It can take weeks to get over the COVID-19 disease; however, some symptoms persist even after the infection has cleared. The continuation of physical, cognitive and psychological problems in COVID-19 patients recovering from the acute phase of the disease is called 'Post-COVID-19 Syndrome'. A good evaluation and treatment is required to prevent these symptoms in individuals with COVID-19.

Telerehabilitation refers to providing rehabilitation services using electronic communication technologies. In the current pandemic process, the use of telerehabilitation has increased all over the world to help patients without compromising the social distance rule. There is no need for protective equipment as there is no physical contact during telerehabilitation sessions. As a result, patient satisfaction and treatment efficiency are increased by enabling more effective and natural human interaction.

In the literature, there are studies examining the effects of telerehabilitation on individuals who have had COVID-19, but studies examining the effects on healthcare workers who have experienced COVID-19 are insufficient. In this study, which is planned to be done, it is aimed to examine the effects of myofascial relaxation technique on pain and other symptoms through telerehabilitation. The aim of the study is to examine the effects of myofascial relaxation technique applied with the telerehabilitation method on pain level, anxiety, depression, sleep, fatigue and kinesiophobia in healthcare workers with and without COVID-19 infection with pain.

ELIGIBILITY:
Inclusion Criteria:

* Pain associated with COVID-19 infection and persistence of this condition after infection
* Presence of non-COVID-19 related pain and no history of COVID-19 infection
* Being a health worker and working actively
* Volunteering

Exclusion Criteria:

* Using psychiatric medication
* Continuing history of active COVID-19 infection

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 2 minutes
  The intensity of pain felt by individuals in their muscles and joints will be evaluated with a visual analog scale. The Visual Analog Scale is scored from 0 to 10. On this scale, "0" indicates no pain, "10" indicates unbearable severity.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 5 minutes
  Sleep quality will be assessed by the Pittsburgh Sleep Quality Index. This questionnaire is a 19-item scale that assesses sleep quality and disturbance over the past month. A total score of less than 5 indicates good sleep quality. A total score greater than 5 indicates that sleep quality is impaired.
Fatigue Severity Scale | 2 minutes
  Fatigue will be evaluated with the Fatigue Severity Scale. The score of the scale, which consists of a total of 9 questions, varies between 9 and 63, while a total score of 36 and above indicates fatigue.
Tampa Scale of Kinesiophobia | 2 minutes
  Tampa Kinesiophobia Scale will be used to assess fear of movement. Individuals get a total score between 17-68. High scores on the scale indicate high kinesiophobia.
The Patient Health Questionnaire-4 | 2 minutes
  Anxiety and depression will be assessed by the Patient Health Questionnaire-4. This questionnaire In the last 2 weeks, the total score in this questionnaire, which consists of 4 questions in total, is between 0-12, and as the scores increase, the psychological distress situation increases.
Modified Borg Dyspnoea Scale | 2 minutes
  The perception of shortness of breath will be measured with the Modified Borg Dyspnoea Scale. Higher scores on this scale indicate increased dyspnea.
Modified Medical Research Council Dyspnea Scale | 2 minutes
  The perception of shortness of breath during activities of daily living was evaluated using the Modified Medical Research Council Dyspnea Scale. Individuals are asked to choose the statement that best describes the severity of dyspnea among 5 statements scored between 0 and 4. High scores indicate an increased level of dyspnea.
Hospital Anxiety and Depression Scale | 2 minutes
  Anxiety and depression levels will be evaluated with the Hospital Anxiety and Depression Scale. There are 14 questions in total in the scale and each question is scored between 0 and 3. While the questions with odd number of questions evaluate anxiety symptoms; Questions with an even number of questions evaluate the symptoms of depression. High scores indicate increased anxiety and depression. While the cut-off point for anxiety is 10; The cut-off point for depression is 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Ceyhun TOPCUOĞLU, Merkez, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No